CLINICAL TRIAL: NCT00103649
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, 18-Month Study of the Efficacy of Xaliproden in Patients With Mild-to-Moderate Dementia of the Alzheimer's Type
Brief Title: 18-Month Study of the Efficacy of Xaliproden (SR57746A) in Patients With Mild-to-Moderate Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC2946; SR57746
Record Dates: First submitted 2005-02-11; First posted 2005-02-14 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — xaliproden

INTERVENTIONS:
Drug: xaliproden (SR57746A)

SUMMARY:
The purpose of this study is to assess xaliproden's potential capacity of slowing the deterioration of cognitive and global functions in patients with mild to moderate Alzheimer's disease. The patients participating in this study will take orally once daily xaliproden or placebo (inactive substance pill).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease using NINCDS-ADRDA criteria

  * Mild to moderate degree of severity of dementia as assessed by the Mini-Mental State Examination score of 16 to 26 (inclusive)
  * Potential participant may be treated with conventional Alzheimer's disease therapy and must be on stable dose for at least 6 months prior to the randomization and during the entire study period
  * Potential participant must have a reliable caregiver and must be living in a community or in an assisted living facility
  * Mother tongue is English, Spanish or French (oral and written fluency)
  * Signed informed consent from potential participant or legal representative and identified caregiver

Exclusion Criteria:

* Potential participant with any other cause of dementia.
* Potential participant with serious health problems other than Alzheimer's disease
* Use of an investigational drug within two months prior to randomization or during this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1306 (Actual)
Dates: Start 2003-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease assessment scale-cognitive, clinical dementia rating sum of boxes.

SECONDARY OUTCOMES:
Mini-Mental State Examination, Alzheimer's Disease assessment scale-activities of daily life.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (120):
- United States (97):
  - UAB Memory Disorders Clinic, Birmingham, Alabama
  - Barrow Neurology Clinics, Phoenix, Arizona
  - PsyPharma Clinical Research, Inc., Phoenix, Arizona
  - Radiant Research, Scottsdale, Arizona
  - Anaheim Research Center, Anaheim, California
  - Margolin Brain Institute, Fresno, California
  - Coordinated Clinical Research, La Jolla, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pharmacology Research Institute, Northridge, California
  - Pharmacology Research Institute, Riverside, California
  - Pacific Research Network, San Diego, California
  - California Neuroscience Research Medical Group, Sherman Oaks, California
  - Pacific Research Network, Vista, California
  - Radiant Research, Denver, Colorado
  - Associated Neurologist, Danbury, Connecticut
  - Geriatric and Adult Psychiatry, LLC, Hamden, Connecticut
  - Yale University School of Medicine AD Research Unit, New Haven, Connecticut
  - Healthcore, Newark, Delaware
  - Neurology Associates, PA, Wilmington, Delaware
  - Atlantic Institute of Clinical Research, Daytona Beach, Florida
  - Berma Research Group, Hialeah, Florida
  - Miami Research Associates, Miami, Florida
  - Baumel-Eisner Neuromedical Institute in Miami Beach, Miami, Florida
  - Baumel-Eisner Neuromedical Institute, Miami, Florida
  - Anchor Research Center, Naples, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Neurology Clinical Research, Inc., Plantation, Florida
  - CNS Clinical Trials, St. Petersburg, Florida
  - Baumel-Eisner Neuromedical Institute in Miami Beach, Tamarac, Florida
  - Meridien Research, Tampa, Florida
  - Suncoast Gerontology Center USF, Tampa, Florida
  - Radiant Research, Marietta, Georgia
  - Southeastern Geriatric Healthcare, Snellville, Georgia
  - Chicago Center for Clinical Research, Chicago, Illinois
  - Radiant Research Center, Hoffman Estates, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Ruan Neurology, Des Moines, Iowa
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Louisiana Research Associates, New Orleans, Louisiana
  - J. Gary Booker MD, Shreveport, Louisiana
  - Clinical Insights, Glen Burnie, Maryland
  - Summit Research Network Michigan, Inc., Okemos, Michigan
  - Pivotal Research Centers, Detroit Office, Royal Oak, Michigan
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Radiant Research, Las Vegas, Nevada
  - ClinSearch, Inc., Kenilworth, New Jersey
  - The Neuroscience Center of Northern New Jersey, Morristown, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Neurology Group of Bergen County, Ridgewood, New Jersey
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Neurological Association of Albany P.C., Albany, New York
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Parker Jewish Institute for Healthcare and Rehabilitation, Hyde Park, New York
  - Neurobehavioral Research, Inc., Lawrence, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - Behavioral Medical Research of Staten Island, New York, New York
  - Global Research and Consulting, Olean, New York
  - Duke University Medical Center (DUMC) - Dept. of Psychiatry, Durham, North Carolina
  - MedARK Clinical Research, Morganton, North Carolina
  - Piedmont Medical Research Assoc, Inc., Winston-Salem, North Carolina
  - DayStar Clinical Research, Inc., Akron, Ohio
  - North East Ohio Health Services, Beachwood, Ohio
  - Valley Medical Primary Care, Centerville, Ohio
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Triphase Research, Ltd., Franklin, Ohio
  - TriPhase Research, Franklin, Ohio
  - Neurology and Neuroscience Center of Ohio, Toledo, Ohio
  - Radiant Research Eugene, Eugene, Oregon
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - Summit Research Network Inc, Portland, Oregon
  - Coatesville VA Medical Center, Coatesville, Pennsylvania
  - Pearl Clinical Research, Norristown, Pennsylvania
  - Memory Disorders Clinic, Philadelphia, Pennsylvania
  - Radiant Research, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, Pittsburgh, Pennsylvania
  - JRMC Clinical Trials Center, Pittsburgh, Pennsylvania
  - RI Mood and Memory, East Providence, Rhode Island
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Avera Research Institute, Sioux Falls, South Dakota
  - CNS Healthcare, Memphis, Tennessee
  - Vanderbilt University Medical Center - Geriatric Psychiatry, Nashville, Tennessee
  - University of Texas - Southwestern Medical Center at Dallas, Dallas, Texas
  - Houston Sleep Center, Houston, Texas
  - AD Research Center, Houston, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - North Texas Neurology Research, Wichita Falls, Texas
  - Radiant Research SLC, Salt Lake City, Utah
  - The Memory Clinic, Bennington, Vermont
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Internal Medicine Northwest, Tacoma, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Dean Foundation, Middleton, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - IPC Research, Waukesha, Wisconsin
- Canada (23):
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - Kelowna, British Columbia
  - Medical Arts Health Research Group, Penticton, British Columbia
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Davidson Memory Clinic, Moncton, New Brunswick
  - St. Joseph's Hospital, Saint John, New Brunswick
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - St. Joseph's Health Care, London, Ontario
  - Parkwood Hospital - Geriatric Medicine, London, Ontario
  - Parkinson's & Neurodegenerative Disorders, Ottawa, Ontario
  - S.C.O. Health Centre, Ottawa, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - University Health Network - The Toronto, Toronto, Ontario
  - NeuroSearch Developments Inc, Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
  - Centre de Hospitalier Affilie, Québec, Quebec
  - Quebec Memory & Motor Skills Disorders, Québec, Quebec
  - Institut Universitaire de Geriatrie de Sherbrooke, Sherbrooke, Quebec
  - Douglas Hospital Research Centre, Verdun, Quebec
  - Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com